CLINICAL TRIAL: NCT05661006
Title: Study of the Efficiency of the Innovative Food Supplement in Improving Nutritional Status of Elderly Adults
Brief Title: ETOL-Elderly Study of the Efficiency of the Innovative Food Supplement in Elderly Adults
Acronym: ETOL-Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: Vizera d.o.o. (Industry); Frutarom Etol d.o.o. (Industry); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020/1-ET-SK
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Vitamin d Deficiency; Vitamin B 12 Deficiency; Protein Deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Vitamin B 12 Deficiency; Protein Deficiency

STUDY DESIGN:
Intervention Model Description: This was a randomized, parallel, double-blind, placebo-controlled study included healthy elderly adults (age > 65 years) who tested study products. On screening visit, participants underwent measuring of body weight & height, and blood collection for measuring S-25-OH-VitD, S-VitB12, S-protein, S-albumin, S-CRP. Duration of study intervention for individual participant 56 ± 3 days, with one week pre-intervention monitoring of food intake (3x 24-h dietary records). On day 1 of the intervention period, participants were randomised in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized on the first day of Visit 1 using simple randomisation using ratio 1:1 between test and placebo group.
  After the general subject's health is checked (vital signs), subjects will be assigned Subject Number, which will be pre-randomised to correspond with one of interventions (test group, placebo group).
  To assure double blind approach, study products will be packed in neutral packaging, and pre-labelled with Subject Number (S-XXX) and instructions for use. Selected site will be provided enough product i.e. subject boxes with corresponding Subject Number to cover initially planned number of included subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Subjects taking control product
  Interventions: Dietary Supplement: Use of placebo food supplement
- Active group (Experimental): Subjects taking active product
  Interventions: Dietary Supplement: Use of food supplement

INTERVENTIONS:
Dietary Supplement: Use of food supplement — On day 1 subjects start with intervention on prearranged day. First dosage of test product is consumed during day 1 between regular meals (not as meal substitute).
  In the following days: continuation of consumption of test product once per day until end of the intervention. Subjects are recording daily consumption of the product. Intervention diet recording during last week of intervention (days 49-56): 3x24h dietary records (two days during weekday, one weekend day).
  Intervention end on day 56 ±3 (fasted condition):
  Measuring S-25-OH-VitD, S-VitB12, S-protein, S-albumin, S-CRP Measuring body weight & height Collecting data regarding the palatability of the product
  Arms: Active group
Dietary Supplement: Use of placebo food supplement — On day 1 subjects start with intervention on prearranged day. First dosage of test product is consumed during day 1 between regular meals (not as meal substitute). In the following days: continuation of consumption of test product once per day until end
  Arms: Control group

SUMMARY:
The aim of this pilot study is to conduct a study on geriatric population in Slovenia (non-users of dietary supplements/medicines with vitamine D, vitamin B12 and protein) and assess deficiency of selected nutrients, and to investigate the efficiency of the innovative food supplement prototype in improving nutritional status of elderly adults.

DETAILED DESCRIPTION:
The main objective is to show that in the geriatric population regular use of investigation food supplement would improve nutritional status. The study should provide answers to the following main questions: (1) Is regular use of investigated product beneficial for improving serum vitamin D levels in elderly population? (2) Is regular use of investigated product beneficial for increasing daily protein intake in elderly population? (3) Is regular use of investigated product beneficial for improving vitamin B12 status in elderly population?

ELIGIBILITY:
Inclusion criteria:

* Subject Informed consent form (ICF) is singed
* Aged at least 65 at the time of the signature of ICF
* A body mass index lower than 32 kg/m2
* Willing to avoid a consumption supplementation with protein, vitamin D and vitamin B12 during the study
* Willing to follow all study procedures, including attending all site visits (including blood sampling) and keeping a diary for using the product and six 24-hour dietary records (3x pre-intervention, 3x during last week of the intervention)

Exclusion criteria:

* Medical treatment with Vitamin D and/or Vitamin B12
* Supplementation with protein, vitamin D and/or vitamin B12 during least 2 months
* Known drug and/or alcohol abuse
* Known lactose/gluten intolerances/food allergies
* Inadequate veins (in the opinion of the investigator) or known contraindication for venous blood withdrawal
* Have chronic bowel disease (ulcerative colitis, Chron's disease, stomach or duodenal ulcer, chronic inflammation of the stomach or duodenum)
* Have acute gastrointestinal infection with vomiting and / or diarrhea
* Have planned general anaesthesia or colonoscopy at the time of the study
* Have malabsorption syndrome
* Less than 5 years after treatment for gastrointestinal cancer (stomach, duodenum or colon)
* Have stomach or bowel resection
* Do not have neat and functional teeth
* Take regular or occasional laxative products
* Use antacids (Rupurut / Rutacid / Talcit)
* Mental incapacity that precludes adequate understanding or cooperation
* Participation in another investigational study

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Change in serum vitamin D levels will be determined | 56 days
  Serum level of 25-OH-vitamin D will be measured before and after the intervention for each individual.

SECONDARY OUTCOMES:
Change in dietary protein intake will be determined | 56 days
  Dietary protein intake will be estimated before and after the intervention for each individual, using 3x24h food records.
Change in serum vitamin B12 levels will be determined | 56 days
  Serum level of vitamin B12 will be measured before and after the intervention for each individual.
Malnutrition at baseline | baseline
  Risks for malnutritition at baseline will be assessed using dietary records (3x24h food record: energy, protein and plasma concentration of 25-OH-D and vitamin B12.

CONTACTS AND LOCATIONS:
Overall Officials: Mojca Miholič, MD, Principal Investigator — Researcher
Locations (1):
- VIZERA, Trzin, Slovenia

IPD SHARING:
Plan to Share IPD: No